CLINICAL TRIAL: NCT02711930
Title: Effect of Prone Positioning on Intra-ocular Pressure in Patients With Acute Respiratory Distress Syndrome (ARDS)
Brief Title: Effect of Prone Positioning on Intra-ocular Pressure in ARDS Patients
Status: Completed | Type: Observational
Sponsor: Sanjay Gandhi Postgraduate Institute of Medical Sciences (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2016-55-DM-EXP
Record Dates: First submitted 2016-03-08; First posted 2016-03-17 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: intra-ocular pressure; prone ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Acute respiratory distress syndrome (ARDS) commonly complicates acute illness in intensive care units (ICU). This syndrome is associated with high morbidity and mortality. In management of ARDS patients, lung protective ventilation and prone ventilation are key strategies which have shown survival benefits in recent years and now become standard part of care in these patient. Prone positioning used for surgeries in operation room has been reported with ocular complications, of which vision loss is one of the devastating complications. There is scarcity of literature on effect of prone positioning on intra-ocular pressure (IOP) in critically ill patients. The purpose of our study is to evaluate the effect of prone position on IOP in critically ill patients and follow up for other ocular complication among survivors.

DETAILED DESCRIPTION:
Introduction and rationale of the study:

Acute respiratory distress syndrome (ARDS) commonly complicates acute illness in intensive care units (ICU). This syndrome is associated with high morbidity and mortality. In management of ARDS patients, lung protective ventilation and prone ventilation are key strategies which have shown survival benefits in recent years and now become standard part of care in these patient.

Prone positioning used for surgeries in operation room has been reported with ocular complications, of which vision loss is one of the devastating complications. Multiple risk factors are reported but orbital compression during prone positioning, excess intravenous fluids, hypotension and duration of prone positioning were the predominant factors. Perioperatively patients, who underwent prone positioning for surgeries can be followed up for symptoms of any complications after the surgery, but this follow up for symptoms is difficult in intensive care units as most of the patients after prone ventilation, will not be able to communicate. The hours of prone ventilation are nearly 3-4 times more, when compared intra-operatively which can definitely increase intra-ocular pressure(IOP) significantly. Most of the patients will be hemodynamically unstable on vasopressor supports, unlike intra-operatively, which can significantly affect ocular perfusion pressure (mean arterial pressure - intra-ocular pressure), making ICU patients with definitely high risk for ocular complication. The purpose of our study is to evaluate the effect of prone position on IOP in critically ill patients and follow up for other ocular complication among survivors.

Tonometry guided IOP measurement is one of the commonly used modality to assess IOP. It has been used in assessing IOP in prone position in awake volunteers with documented increase in IOP within few hours of prone positioning on operating tables It has been studied under anesthesia with elevated IOP and significantly increased IOP in the dependent eye.

Primary objective:

• To evaluate the effect of prone positioning on intraocular pressure (IOP) in critically ill patients with acute respiratory distress syndrome.

Secondary objectives:

• To follow up survivors for detailed ophthalmological examination of anterior and posterior segment of both eye.

Work plane methodology:

Prospective observational study will be conducted in Department of Critical Care Medicine, SGPGIMS, Lucknow after Institutional Ethics Committee approval. Consent from the patient's family member will be obtained.

All adult patients with ARDS who are planned for prone ventilation, as decided by the treating physician, will be screened for inclusion in this study. As a part of standard treatment for ARDS, all patients will be receiving lung protective ventilation strategies as per ARDS net protocol with appropriate sedation and paralysis, and also these patients will have relevant invasive and non-invasive vitals monitoring as per ICU protocol. All IOP measurements will be taken by same investigator throughout the study, who will be trained to monitor IOP in ten patients under direct supervision of an experienced ophthalmologist. In studied patients, baseline readings of IOP will be measured by tonometry device before prone positioning in 30-45 degree head end elevation (T1). Next reading of IOP will be measured (T2), 5 minutes after supine position, i.e. during preparation for turning the patient prone. Then, patients will be proned with adequate precautions to avoid ocular compression and rest of the body supported with adequate thoraco-pelvic supports. Duration of prone ventilation will be decided by treating physician. The next IOP will be measured in non-dependent eye at 10 minutes (T3) and 30 minutes (T4) of prone position; and just before making the patient supine (T5). After completion of prone position session, IOP will be measured again in both eyes at 5 minutes after turning the patient in supine without head end elevation (T6), then followed by measurement at 10 minutes (T7), 15 minutes (T8) and at 30 minutes (T9). Last 3 measurements i.e. T7, T8 and T9 will be done in 30-45 degree head end elevation. All IOP values will be recorded as a mean of three readings at each pre-defined time, in both eyes of the patient. Monitored vitals with relevant clinical data will be noted. Patient will be followed till ICU discharge. Detailed ophthalmic examination for anterior segment (which includes IOP measurement); and posterior segment of both eyes will be done in survivors at time of ICU discharge as well as at 1 month and at 3 months, in follow up.

Sample size calculation:Sample size was calculated using minimum 95% confidence interval and 95% power of the study for one group in which observation will be taken in six times as repeated design. Assuming 0.28 standard deviation of the effect size of the mean difference, calculated sample size came out to be 23. Finally for this study, sample size has been taken 25. PASS-8 (Power and sample size) software version 8 have been used to calculate sample size.

Data Collection: Demographic and relevant clinical characteristics of all included patients will be collected on structured proforma. ICU prognostication scores, i.e., Acute Physiologic and Chronic Health Evaluation (APACHE) II score and Sequential Organ Dysfunction Assessment (SOFA) will also be recorded. Duration of prone ventilation as well as position of head (right or left side turn) will also be noted down. IOP will be measured for both eyes at pre-defined time intervals. Detailed ophthalmic examination findings will be collected among survivors at time of ICU discharge and after 3 months in follow up.

Intervention: Nil. All patients will be managed as per the ICU treating team's decision

ELIGIBILITY:
Inclusion Criteria:

• Adult (age >18 years) patients with ARDS requiring prone ventilation

Exclusion Criteria:

* Patient with age <18 years
* Clinical conditions with suspected raised intra-cranial pressure (ICP)
* Previous eye trauma or disease or surgery
* Patients with family history of glaucoma or history of pain and redness of eye (obtained from patient's family)
* Any prone positioning of less than 6 hours duration (planned or unplanned)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having acute respiratory distress syndrome and requiring prone ventilation during ICU stay.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2016-05-03 (Actual); Primary Completion 2017-07-24 (Actual); Study Completion 2017-10-24 (Actual)

PRIMARY OUTCOMES:
To study percentage change in intra-ocular pressure due to prone positioning in patients with ARDS. | Baseline (pre-prone) and after termination of prone position (post-prone) at 5, 10, 15 and 30 minutes.
  The investigators will study percentage change in intra-ocular pressure due to prone positioning in patients with ARDS.

SECONDARY OUTCOMES:
Ophthalmic examination for anterior segment and posterior segment of both eyes will be done in survivors. | Before discharge from intensive care unit, and after that at 1 month and at 3 months, in follow up.
  The investigators will do ophthalmic examination for anterior segment and posterior segment of both eyes among survivors.

CONTACTS AND LOCATIONS:
Overall Officials: Mohan Gurjar, MD, PDCC, Principal Investigator — Sanjay Gandhi Postgraduate Institute of Medical Sciences
Locations (1):
- Department of Critical Care Medicine, SGPGIMS, Lucknow, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Saran S, Gurjar M, Kanaujia V, Ghosh PS, Gupta A, Mishra P, et. al. Effect of Prone Positioning on Intraocular Pressure in Patients With Acute Respiratory Distress Syndrome. Crit Care Med. 2019 Sep;47(9):e761-e766. PMID: 31305498 — https://www.ncbi.nlm.nih.gov/pubmed/31305498